CLINICAL TRIAL: NCT04166175
Title: Treatment of Chronic Anal Fissure, Lateral Internal Sphincterotomy Versus Local Injection of High Dose Botulinum Toxin: A Randomized Clinical Trial
Brief Title: High Dose Multiple Site Injection of Botox Versus Lateral Sphincterotomy in Chronic Analfissure
Acronym: professor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Nour Abdellatif, Assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anal sphincterotomy or botox
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Chronic Anal Fissure
MeSH Terms: interventions — Botulinum Toxins, Type A; Lateral Internal Sphincterotomy

STUDY DESIGN:
Intervention Model Description: two groups of patients randomly allocated group1 the botox group received 80 IU botox injection and group 2 under went lateral internal sphincterotomy
Who Masked: Participant
Masking Description: participant don't know the procedure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 botox group (Active Comparator): 48 patients subjected to 80 IU botox injection under GAin lithotomy position in the 5,7,11, and 1 O'clock positions
  Interventions: Procedure: botox injection in intersphincteric space
- group 2 lateral sphincterotomy group (Active Comparator): 48 patients subjected to lateral internal sphincterotomy under GAin lithotomy position
  Interventions: Procedure: lateral internal sphincterotomy

INTERVENTIONS:
Procedure: botox injection in intersphincteric space — injection of 80 IU of botox in the intersphincteric space in 5,7,11 and 1 O'clock position
  Arms: group 1 botox group
Procedure: lateral internal sphincterotomy — lateral internal sphincterotomy under GA in lithotomy position
  Arms: group 2 lateral sphincterotomy group

SUMMARY:
comparison between the effect of lateral sphincterotomy against high dose botox injection in chronic anal fissure the outcome was healing time, recurrence continence relapse pain pruritus

DETAILED DESCRIPTION:
This randomized comparative clinical trial was carried out over 2 year in the period between January 2018 and December 2019 on total number of 96 patients suffering chronic anal fissure the participants were randomly allocated into two groups each 48 patients ; group (1) the botulinum ( Botox) group, they were subjected to 80 IU Botox injection as an intervention for treatment of chronic anal sphincter, and group 2 the sphincterotomy group, underwent internal sphincterotomy as a surgical intervention for treatment of chronic anal fissure.

The study was approved by the institutional review board and the local ethical committee of our university hospital The condition of the current study is chronic anal fissure defined as the presence of anterior or posterior chronic anal wound with skin tag at its lower end and hypertrophied anal papilla at its upper end with induration around its edges in patients complaining of anal pain, constipation, and/or fresh anal bleeding for at least two months.

Randomization was achieved using computer generated cards. Inclusion criteria; patients suffering chronic anal fissure aged above 16 years old Exclusion criteria; those with previous anal surgery, complicated anal fissure, unfit for surgery, specific disease as Crohn's disease and ulcerative colitis, malignancy, anal fistula or abscess those with systemic disease requiring treatment with calcium channel blockers and /or nitrates Patients of both groups were subjected to thorough history taking, clinical examination, digital rectal examination and anorectal manometry for diagnosis of chronic anal fissure and exclusion of any other anal condition and incontinence, patient signed an informed written consent, routine preoperative investigations performed as usual.

Interventions;

1. Botulinum toxin (Botox) injection; was performed under general anesthesia in the lithotomy position, where 80 IU of Botox was injected in four positions each 20 IU namely in 5, 7, 11, and 1 O'clock positions in the intersphincteric space not deeper than the midpoint of the anal canal.
2. Lateral internal sphincterotomy; was performed under general anesthesia where the lower part of the internal sphincter was cut by electrocautery on the left lateral position to an extent not beyond the proximal end of the fissure, the sentinel pile was also removed.

After the procedure patients were advised for bulking agents, stool softener, and sitz baths The follow up was carried out in the outpatient clinic by the attending surgeon (not a study participant) after 1 week then 1, 2, 3, 6, 9 and 12 months post-procedure.

The primary outcome of the current study is complete healing of the chronic anal fissure, recurrence in the follow up time, and development of incontinence, incontinence is described as in (the Cleveland Clinic Florida-Fecal Incontinence (CCF-FI) scoring system), which contains 5 questions on solid and liquid stool leakage, gas leakage, pad use, and lifestyle restriction. the secondary outcome is postoperative or post-injection pain measured by visual analogue scale (VAS) and the time taken for complete healing of fissure (defined as complete epithelialization of the fissure).

Demographic data, presentation data, follow up data including primary and secondary outcome all collected and analyzed properly using t test, chi square test, and Z test in SPSS program 22 version.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering chronic anal fissure aged above 16 years old

Exclusion Criteria:

* those with previous anal surgery,
* complicated anal fissure,
* unfit for surgery,
* specific disease as Crohn's disease and ulcerative colitis,
* malignancy,
* anal fistula or abscess
* those with systemic disease requiring treatment with calcium channel blockers and /or nitrates

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
complete healing of fissure | 2 months
  complete epithelialization of the floor of the chronic anal wound achieved through clinical examination at follow up visits
loss of anal continence | 1 week
  inability to control stool or flatus measured by modified wexner score questionaire
recurrence | 1 year
  the anal fissure reformed again after complete healing measured by clinical examination

SECONDARY OUTCOMES:
time taken for complete healing | 1 year
  time taken for complete epithelialization of the anal wound measured by clinical examination
post operative pain | 1 month
  pain in the postoperative time measured by visual analogue scale

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig Faculty of Medicine, Zagazig, Sharqya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided